CLINICAL TRIAL: NCT02830152
Title: Prevention of Stroke by Left Atrial Appendage Closure in Atrial Fibrillation Patients After Intracerebral Hemorrhage: A Multicenter Randomized Clinical Trial
Brief Title: Prevention of Stroke by Left Atrial Appendage Closure in Atrial Fibrillation Patients After Intracerebral Hemorrhage
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Per Wester, Principal investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STROKECLOSE
Record Dates: First submitted 2016-06-29; First posted 2016-07-12 (Estimated); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Atrial Fibrillation; Stroke; Intracerebral Hemorrhage
Keywords: Stroke; intracerebral hemorrhage; left atrial appendage occlusion; atrial fibrillation; oral anticoagulation; preventive therapy
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Cerebral Hemorrhage | interventions — Nutrition Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left Atrial Appendage Occlusion (LAAO) (Experimental): The intervention is implantation of Amplatzer Amulet LAAO device within two months after randomization. Device implantation comprises a catheterization procedure using venous access and a transseptal puncture to obtain access to the left atrium (LA). Procedural imaging guidance is left to the physician's discretion and may include several techniques such as angiography/fluoroscopy, transesophageal echocardiography (TEE) and/or intracardiac echocardiography (ICE). Recommended post-implant antithrombotic therapy includes ASA therapy for at least 6 months, which may be combined with clopidogrel for the first 45 days after implantation.
  Interventions: Device: LAAO
- Medical Therapy (Active Comparator): The optimal medical therapy of stroke prevention in non-valvular atrial fibrillation (NVAF) after intracerebral hemorrhage (ICH) is not known. Therefore, it will be left to the discretion of the treating physician to decide if, when, and which pharmacological therapy will be prescribed. Available options include anticoagulation with oral anticoagulation (OAC) or novel oral anticoagulants (NOAC), antiplatelet therapy (including monotherapy and dual antiplatelet therapy) and no pharmacological antithrombotic therapy.
  Interventions: Drug: Medical Therapy

INTERVENTIONS:
Device: LAAO — The left atrial appendage is occluded with the AMPLATZER™ Amulet™ device, which offers a conformable disc and lobe designed for complete occlusion of the left atrial appendage.
  Other Names: AMPLATZER™ Amulet™ (St. Jude Medical)
  Arms: Left Atrial Appendage Occlusion (LAAO)
Drug: Medical Therapy — Available options included in Medical therapy are: anticoagulation with OAC or NOAC, antiplatelet therapy (including monotherapy and dual antiplatelet therapy) and no pharmacological antithrombotic therapy.
  Other Names: Antiplatelet Therapy
  Arms: Medical Therapy

SUMMARY:
Intracerebral hemorrhage (ICH) in patients with non-valvular atrial fibrillation (NVAF) poses a particular dilemma for thromboprophylaxis. Left atrial appendage occlusion (LAAO) is a non-pharmacological approach to prevent cardiac embolism in NVAF. The risk-benefit ratio of LAAO in patients with NVAF after ICH is unknown. The aim of STROKECLOSE is to assess the effect of LAAO to reduce the incidence stroke, bleeding and cardiovascular mortality in patients with NVAF and prior ICH.

DETAILED DESCRIPTION:
Methods/design: A multicenter prospective randomized open-label clinical trial with blinded outcome evaluation (PROBE design) and blinded safety outcome assessment. The active comparison LAAO is tested against medical therapy in a 2:1 stratified randomization.

Study population: Patients should have had an ICH within 12 months prior to enrollment and have NVAF with increased risk of stroke or systemic embolism, as indicated by a CHA2DS2VASc score >2. In total 750 patients will be included. Active enrollment ensues over 3 years followed by 5 years follow-up and a long-term follow-up at 10 years.

Intervention and control: The intervention group will be treated by LAAO, using the Amplatzer Amulet device. Implantation requires a catheterization procedure using venous access and transseptal puncture and is guided by angiography, fluoroscopy and transesophageal echocardiography (TEE) or intracardiac echocardiography (ICE). Recommended post-implant antithrombotic therapy includes aspirin (ASA) therapy for at least 6 months, with or without clopidogrel for the first 45 days after implantation. The control group will receive medical therapy, delivered according to national standards and guidelines at the treating physicians' discretion. This may include oral anticoagulation (OAC) (vitamin-K antagonists, VKA), non-VKA OAC, antiplatelet therapy or no antithrombotic therapy at all.

Main study outcomes: The primary outcome is the composite endpoint of stroke (ischemic and hemorrhagic), systemic embolism, life-threatening or major bleeding and all-cause mortality, assessed over at least two years. Secondary outcome examines various early and late safety outcome parameters.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of paroxysmal, persistent or long-standing NVAF with CHA2DS2VASc score >2.
* Clinical and CT/MRI evidence of ICH within 12 months but not less than 4 weeks prior to enrollment.
* Age > 18 years.
* Signed informed consent.

Exclusion Criteria:

* ICH secondary to vascular malformation or tumors
* Estimated life expectancy of less than 1 year at eligibility assessment
* mRS > 3 at enrollment
* Prior surgical LAA excision
* Planned combined interventional procedures at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of stroke (ischemic or hemorrhagic), systemic embolism, life-threatening or major bleeding and all-cause mortality | up to 5 years after randomization
  This endpoint will be assessed in patients with paroxysmal, persistent or long-standing NVAF and with ICH within 6 months prior to enrollment.
  The effect of LAAO will be compared to medical therapy at the treating physician's discretion as a control.

SECONDARY OUTCOMES:
Number of participants with a device-related complication | up to 45 days after randomization
  A complication related to the presence of the device. Device-related complications include:
  * Device embolization
  * Device erosion
  * Clinically significant device interference with surrounding structures. This includes structures at the implant location (circumflex coronary artery, mitral valve, pulmonary artery, pulmonary vein) or cardiovascular structures in the vicinity of the location to which the device migrated (if applicable).
  * Device thrombus
  * Device fracture
  * Device infection/endocarditis/pericarditis
  * Device perforation/laceration
  * Device allergy
Number of Participants with a device success | up to 45 days after randomization
  Device deployed and implanted in correct position.
Number of Participants with a Technical success | up to 45 days after randomization
  Exclusion of the left atrial appendage (LAA) achieved without device-related complications and no leak >5 mm on color Doppler TEE.
Number of Participants with a Procedural success | up to 45 days after randomization
  Technical success and no procedure-related complications, except uncomplicated device embolization (i.e. device embolization resolved by percutaneous retrieval during the procedure without surgical intervention or damage to surrounding cardiovascular structures).
Number of Participants with Significant peridevice leak | up to 45 days after randomization
  Consistent with the definition of technical success, a significant peridevice leak is defined as a leak shown as a jet >5 mm on color Doppler TEE.
Compare the functional status prior to and post treatment | 24 months after randomization
  The Modified Rankin Scale (mRS) will be used for measuring the Functional status.
Compare the cognitive status prior to and post treatment | 24 months after randomization
  The cognitive status will be assessed by using Montreal Cognitive Assessment (MOCA) and Mini-mental state examination (MMSE)
Compare the neurological status prior to and post treatment | 24 months after randomization
  The National Institutes of Health Stroke Scale (NIHSS) is used to assess the neurological status
Compare the quality of life prior to and post treatment by using EuroQol | 24 months after randomization
  EuroQol assesses health status in terms of five dimension: mobility (walking about); looking after myself; doing usual activities (e.g., going to school, hobbies, sports, playing, doing things with family and friends); having pain or discomfort; and feeling worried, sad, or unhappy. The levels for the dimensions are: 'none/no problems', 'some (problems)', and 'a lot (of problems)'. Higher score represents more problems.
Late safety outcome parameters of LAAO and Medical therapy | up to 10 years after randomization
  Stroke (ischemic or hemorrhagic), systemic embolism, bleeding, all-cause mortality, intracranial hemorrhage, cardiovascular mortality and unplanned hospitalization will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Per Wester, MD, Principal Investigator — Department of Clinical Sciences, Karolinska Institute, Danderyds hospital
Locations (17):
- Denmark (5):
  - Aarhus University Hospital, Aarhus
  - Bispebjerg University Hospital, Bispebjerg
  - Rikshospitalet Glostrup, Glostrup Municipality
  - Herlev sjukhus, Herlev
  - Odenses Universitetssjukhus, Odense
- Finland (5):
  - Helsinki University Hospital, Helsinki
  - North Karelia Central Hospital, Joensuu
  - Kuopio University Hospital, Kuopio
  - Turku University Hospital, Turku
  - Vaasa Centralsjukhus, Vaasa
- Norway (2):
  - Haukeland Universitetssjukhus, Bergen
  - Oslo University Hospital, Oslo
- Sweden (5):
  - Sahlgrenska University Hospital, Gothenburg
  - Universitetssjukhuset Skåne, Lund
  - Universitetssjukhuset, Örebro
  - Danderyd Hospital, Stockholm
  - Akademiska sjukhuset, Uppsala

IPD SHARING:
Plan to Share IPD: Yes
The full study protocol, statistical plan and informed consent form will be publicly available when results are published. Data will be available on patient level; data will be pseudonymized. The full dataset will be available upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting after publication and for 36 months.
Access Criteria: A full description of the intended use of the data must be sent to the corresponding author for review and approval. Participant consent for data sharing is conditioned and new ethics approval may be required.